CLINICAL TRIAL: NCT05446935
Title: Cytoreductive Surgery and Hyperthermic Intrathoracic Chemotherapy for the Treatment of Thymic Epithelial Malignancies With Pleural Spread or Recurrence (CHOICE): a Prospective, Open, Single-arm Study Choice
Brief Title: Intrathoracic Chemotherapy for TETs With Pleural Spread or Recurrence
Acronym: CHOICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2021-703R
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Thymic Epithelial Tumor
Keywords: Hyperthermic Intrathoracic Chemotherapy; Thymic Epithelial Malignancies
MeSH Terms: conditions — Thymic epithelial tumor

STUDY DESIGN:
Intervention Model Description: A Prospective single-arm Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HITOC (Other): HITOC group contains all patients who undergo HIROC in this study.
  Interventions: Procedure: HITOC

INTERVENTIONS:
Procedure: HITOC — Doxorubicin(dose: 25mg/m2) + Cisplatin(dose: 50mg/m2).

SUMMARY:
Hyperthermic intrathoracic chemotherapy (HITOC) offers an additional treatment option for malignant pleural tumors after surgical cytoreduction. Especially it is used to further improve local tumor control in thymic malignancies with pleural spread, who underwent multimodality therapy including surgical resection. A phase II clinical study was conducted to explore the efficacy and safety of surgery followed by HITOC (POD1: DOX, POD2: cisplatin) for thymic epithelial tumors with pleural spread or recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Puncture biopsy, thoracoscopic/mediastinal biopsy, or surgery to confirm pathologically thymic epithelial tumor (TETs)
2. Imaging examination shows TETs with pleural spread or recurrence, and the mediastinal MDT team considers HITOC suitable.
3. Patients with ≥16 and ≤80 years old.
4. ASA I-II.
5. The patients should have no functional disorders in the main organs.
6. There was no history of other malignant carcinomas.
7. The duration from the last chemotherapy was >4 weeks, the duration from the last radiotherapy was >6 weeks, and the duration from the last immunotherapy was >6 weeks.
8. Not allergic to cisplatin or doxorubicin.
9. The patients should be able to understand our research and sign the informed consent.

Exclusion Criteria:

1. Imaging or pathological examination shows TETs without pleural spread or recurrence, or with pericardial dissemination or extrathoracic metastasis.
2. Patients with lymphoid system, neurogenic or reproductive system carcinoma.
3. Patients who have been receiving chemotherapy, radiotherapy, immunotherapy, or targeted therapy.
4. Patients with myasthenia gravis in unstable or acute exacerbation stage.
5. The patients have been proven history of congestive heart failure, angina without good control with medicine; ECG-proved penetrating myocardial infarction; hypertension with bad control; valvulopathy with clinical significance; arrhythmia with high risk and out of control.
6. The patients have the severe systematic intercurrent disease, such as active infection or poorly controlled diabetes; coagulation disorders; hemorrhagic tendency or under-treatment of thrombolysis or anticoagulant therapy.
7. Female who is positive for a serum pregnancy test or during lactation period.
8. The patients have a history of organ transplantation (including autologous bone marrow transplantation and peripheral stem cell transplantation.
9. The patients have a history of peripheral nerve system disorders, obvious mental disorders, or central nerve system disorders.
10. The patients attend other clinical trials.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative hospital stay | Up to the date of meeting the criteria of hospital discharge since the data of surgery, up to 1 month
  Postoperative hospital stay is the duration for every enrolled patient until the date of meeting the criteria of hospital discharge since the date of surgery.
  The criteria of hospital discharge were defined as with the volume of postoperative drainage < 200 ml/day, a normal chest X-ray, and good physical condition.
treatment-related adverse events and complications | Up to the date of meeting the criteria of hospital discharge since the data of surgery, up to 1 month
  Number and severity of adverse events that are related to the treatment of each patient. Postoperative treatment-related complications were assessed by the Clavien-Dindo Classification. Treatment-related adverse events as assessed by CTCAE v5.0.
EORTC QLQ-C30 score for overall quality of life | Up to the end of follow-up since the date of randomization, up to 6 months.
  Overall quality of life is respectively evaluated at randomization and 1 month, 3 month, 6 month after surgery among patients by using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 Scale (EORTC QLQ-C30) (V3.0).
  The minimum value of EORTC QLQ-C30 score was 0， and the maximum was 100. Zero indicates the worst quality of life, while 100 represents the best quality of life.

SECONDARY OUTCOMES:
Visual Analog Scales scores for postoperative pain | from 0 to 72 hours after surgery
  the cumulative daily pain score at rest using VAS from postoperative 0 to 72 hours. The minimum value of the VAS score was 0，and the maximum was 10. Zero indicates the least painful, while 1 represents the worst. The smaller (larger) cumulative daily pain score represents the less (more) pain.
Volume of postoperative drainage | Up to the date of removal of drainage equipment since the data of completion of surgery, up to 7 days
  The volume of postoperative drainage of the patient was the sum of his daily drainage volume after the surgery. The types of drainage equipment include the thorax close drainage equipment and the unidirectional negative-pressure drainage ball.
Progression-free survival (PFS) | Through study completion, an average of 5 year
  the duration from the date of S-HITOC to the date of the first progression. Disease progression is defined as locoregional (anterior mediastinal area, lung, pericardiac metastasis or pleural progression) or metastatic (supraclavicular lymph nodes or distant organs).
Overall survival (OS) | Through study completion, an average of 5 year
  the duration from the date of S-HITOC to the date of the death.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

REFERENCES:
- [Derived] Wang S, Yang X, Jiang J, Liang F, Zheng Y, Ao Y, Gao J, Wang H, Tan L, Ding J. Cytoreductive surgery and hyperthermic intrathoracic chemotherapy in thymic epithelial tumors with pleural spread or recurrence: a prospective, single-arm, phase II study. Nat Commun. 2025 Jun 4;16(1):5175. doi: 10.1038/s41467-025-60386-0. PMID 40467556
- [Derived] Yang X, Wang S, Jiang J, Lin M, Gao J, Ding J, Tan L. Cytoreductive surgery combined with hyperthermic intrathoracic chemotherapy for the treatment of thymic epithelial malignancies with pleural spread or recurrence (CHOICE): a study protocol for a prospective, open, single-arm study. J Thorac Dis. 2024 Jan 30;16(1):760-767. doi: 10.21037/jtd-23-759. Epub 2023 Dec 25. PMID 38410567